CLINICAL TRIAL: NCT07312032
Title: The Effects of Footplate Stiffness on Foot Loading Within Carbon Fiber Custom Dynamic Orthoses
Acronym: CDOCFPlate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Wilken (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Jason Wilken, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202507360; 202507360 (Other: University of Iowa)
Record Dates: First submitted 2025-12-29; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Trauma Injury
Keywords: carbon fiber; traumatic injury; ankle foot orthosis
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: In this study participants will walk without an orthosis (NoCDO) and with a generic sized CDO with three different levels of footplate stiffness at a controlled speed (CDO, 1CFPlate, 2CFPlate). Testing order of the CDO conditions will be randomized to prevent influence of testing order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- NoCDO (No Intervention): Participants will complete study activities without a CDO
- CDO (Experimental): Participants will complete study activities while wearing a CDO with standard footplate stiffness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis
- 1CFPlate (Experimental): Participants will complete study activities while wearing a CDO with standard footplate stiffness and one additional carbon fiber footplate to increase footplate stiffness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis; Device: Carbon Fiber Footplate
- 2CFPlate (Experimental): Participants will complete study activities while wearing a CDO with standard footplate stiffness and two additional carbon fiber footplates to increase footplate stiffness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis; Device: Carbon Fiber Footplate

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis — The carbon fiber custom dynamic orthosis (CDO) used in this study will consist of a semi-rigid carbon fiber footplate, a carbon fiber posterior strut, and a proximal cuff that wraps around the leg below the knee.
  Other Names: ankle foot orthosis
  Arms: 1CFPlate; 2CFPlate; CDO
Device: Carbon Fiber Footplate — One or two additional full-length carbon fiber footplates will be placed under the CDO footplate to increase the effective footplate stiffness
  Arms: 1CFPlate; 2CFPlate

SUMMARY:
Carbon fiber custom dynamic orthoses (CDOs) improve function, reduce pain, and offload the foot and ankle. CDOs include a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that bends to store and return energy, and a semi-rigid carbon fiber footplate. The purpose of this study is to determine the effect of CDO use and CDO footplate stiffness on foot loading, limb mechanics, pain, and comfort.

DETAILED DESCRIPTION:
Carbon fiber custom dynamic orthoses (CDOs) have been used to improve function, reduce pain, and offload the foot and ankle for individuals with a number of conditions affecting the lower extremity.[1-3] CDOs consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that bends to store and return energy during mid to late stance, a semi-rigid carbon fiber footplate, and, in some cases, a foam heel wedge placed in the shoe. Studies have previously investigated the effects of design characteristics on gait biomechanics and foot loading, however, the effect of foot plate stiffness on resulting foot loading is unknown.

The purpose of this study is to determine the effect of CDO use and CDO footplate stiffness on foot loading, limb mechanics, pain, and comfort. In this study, forces acting under the foot will be measured using wireless Loadsol insoles (Novel GMBH, St. Paul, MN) and limb mechanics will be measured using motion capture cameras and force plates as participants walk without an orthosis (NoCDO), with a CDO, and with a CDO plus added carbon fiber stiffening inserts (1/2) at a controlled walking speed. Participants will be provided a heel lift for the contralateral limb to prevent leg length discrepancies during walking if necessary. After walking in each condition, participants will complete questionnaires concerning pain and orthosis comfort.

ELIGIBILITY:
Inclusion Criteria

* Between the ages of 18 and 65
* Healthy without current complaint of lower extremity pain, spine pain, open wounds or active infections, or medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Able to hop without pain
* Able to perform a full squat without pain
* Ability to read and write in English and provide written informed consent
* Ability to fit in a generic sized CDO

Exclusion Criteria

* Diagnosed with a moderate or severe brain injury
* Lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Injuries that would limit performance in this study
* Diagnosed with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* Require use of an assistive device
* Unhealed wounds (cuts/abrasions) that would prevent AFO use
* BMI > 40
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Peak Forefoot Force | Baseline
  Plantar forces (N) will be measured across the forefoot (distal 40% of sensor).
Forefoot Force Impulse | Baseline
  Plantar force impulse (Ns) across the forefoot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase.
Peak Hindfoot Force | Baseline
  Plantar forces (N) will be measured across the hindfoot (proximal 30% sensor).
Hindfoot Force Impulse | Baseline
  Plantar force impulse (Ns) across the hindfoot (proximal 30% sensor) will be calculated using the integral of the force over the stance phase.
Peak Ankle Power | Baseline
  Peak sagittal plane ankle push-off power (W/kg) during gait.

SECONDARY OUTCOMES:
Peak Midfoot Force | Baseline
  Plantar forces (N) will be measured across the midfoot (middle 30% of sensor).
Midfoot Force Impulse | Baseline
  Plantar force impulse (Ns) across the midfoot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase.
Peak Total Foot Force | Baseline
  Plantar forces (N) will be measured across the total foot (100% of sensors).
Total Foot Force Impulse | Baseline
  Plantar force impulse (Ns) across the total foot (100% of sensors) will be calculated using the integral of the force over the stance phase.
Peak Ankle Dorsiflexion | Baseline
  Peak ankle dorsiflexion (degrees) during gait.
Peak Ankle Plantarflexion | Baseline
  Peak ankle plantarflexion (degrees) during gait.
Ankle Range of Motion | Baseline
  Range of ankle motion (degrees) during gait.
Peak Ankle Dorsiflexion Moment | Baseline
  Peak ankle dorsiflexion moment (Nm/kg) during gait.
Peak Ankle Plantarflexion Moment | Baseline
  Peak ankle plantarflexion moment (Nm/kg) during gait.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10= most comfortable

OTHER OUTCOMES:
Modified Socket Comfort Score (Smoothness) | Baseline
  Smoothness scores range from 0 = least smooth to 10 = most smooth

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No